CLINICAL TRIAL: NCT03639935
Title: Phase II Multi-Center Study of PARP Inhibitor Rucaparib in Combination With Anti-PD-1 Antibody Nivolumab in Patients With Advanced or Metastatic Biliary Tract Cancer Following Platinum Therapy
Brief Title: Rucaparib in Combination With Nivolumab in Patients With Advanced or Metastatic Biliary Tract Cancer Following Platinum Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.044; HUM00142974 (Other: University of Michigan)
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Cancer
Keywords: Metastatic; Platinum; Rucaparib; Nivolumab; PARP Inhibitor; Anti-PD-1 Antibody
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasm Metastasis | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rucaparib and Nivolumab (Experimental): Rucaparib 600 mg PO BID days 1-28 Nivolumab 240 mg IV days 1 and 15
  Interventions: Drug: Rucaparib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rucaparib — Rucaparib 600 mg PO BID days 1-28
Drug: Nivolumab — Nivolumab 240 mg IV days 1 and 15

SUMMARY:
Investigators hypothesize that following first-line platinum based chemotherapy, rucaparib in combination with nivolumab, will improve progression-free survival and overall survival in BTC patients.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a pathologically confirmed adenocarcinoma of the biliary tract (intra-hepatic, extra-hepatic (hilar, distal) or gall bladder) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed histology are excluded.
* Patients must have received 1st line platinum-based systemic chemotherapy for advanced BTC for 4-6 months without radiologic or clinical progression. Last systemic infusion of 1st line platinum-based therapy may not be more than 4 weeks from study informed consent. Prior peri-operative chemotherapy is permitted provided it was completed > 6 months from start of platinum-based therapy for advanced disease.
* Prior surgical resection, radiation, chemoembolization, radioembolization or other local ablative therapies are permitted if completed > 4 weeks prior to enrollment AND if patient has recovered to < 1 grade 1 toxicity.
* Patients must have measurable disease (as per RECISTv1.1) in at least one site not previously treated with radiation or liver directed therapy (including bland, chemo- or radio-embolization, or ablation) either within the liver or in a metastatic site unless the patient has had complete response to 1st line platinum-based therapy.
* Age≥18 years
* Child-Pugh score of A or B7 (Scoring system used to assess the prognosis of chronic liver disease, mainly cirrhosis)
* ECOG performance status of 0-1 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.)
* Ability to understand and willingness to sign IRB-approved informed consent
* Available archived tissue (FFPE block or 20 unstained slides from prior core biopsy or surgery)
* Must be able to tolerate CT and/or MRI with contrast
* Adequate organ function obtained ≤ 2 weeks prior to registration

Exclusion Criteria

* Diagnosis of immunodeficiency, or received systemic steroid therapy, or any other form of immunosuppressive therapy within 14 days prior to trial treatment. Short bursts of steroids of 5-7 days (for COPD exacerbation or other similar indication) are allowed.
* Prior history of solid organ transplantation or brain metastasis (unless treated and stable)
* Patients may not have undergone a major surgical procedure < 4 weeks prior to registration
* Active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. Patients with history of malignancy are eligible provided primary treatment of that cancer was completed > 1 year prior to registration and the patient is free of clinical or radiologic evidence of recurrent or progressive malignancy.
* Ongoing active, uncontrolled infections (afebrile for > 48 hours off antibiotics)
* Have received a live vaccine within 30 days of planned start of the study therapy
* Have a psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements
* Pregnant or breastfeeding since rucaparib and/or nivolumab may harm the fetus or child. All females of childbearing potential (not surgically sterilized and between menarche and 1-year post menopause) must have a blood or urine test to rule out pregnancy within 2 weeks prior to registration.
* Women of child-bearing potential and men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 6 months (for women) and 7 months (for men) following completion of study therapy
* Participants with an active, known or suspected autoimmune disease which may affect vital organ function, or has/may require systemic immunosuppressive therapy for management. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Patients may not have previously received anti PD1/PDL1 antibodies or PARP inhibitor for treatment of this cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MBBS, MS, Principal Investigator — Rogel Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rogel Cancer Center, Ann Arbor, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results published in peer reviewed research articles, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data is for meta-analysis, and has been approved by an independent review committee identified for this purpose. Proposals should be directed to vsahai@umich.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled, but never treated, as they did not meet lab requirements on C1D1
Period: Overall Study
Arm/Group | Rucaparib and Nivolumab
Started | 31
Completed | 27
Not Completed | 4
Not completed — Death | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Without Radiological or Clinical Progression at 4 Months
Description: Progressive disease is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions (with a minimum absolute increase of 5 mm), taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
  A clinical decision of progression by the site investigator will be based on the subject's overall clinical condition, including performance status, clinical symptoms, and laboratory data.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
percentage of participants | 54.8 [36 to 72.7]

2. Secondary Outcome: The Proportion of Patients That Respond to Treatment
Description: The proportion of patients that display a partial response (PR) or complete response (CR) to treatment.
  Partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
  Complete response is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
Time Frame: up 2 years after starting treatment, average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
Participants | 2

3. Secondary Outcome: Progression Free Survival (PFS) Time as Measured From Treatment Start
Description: Progressive disease is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions (with a minimum absolute increase of 5 mm), taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
months | 4.6 [3.7 to 6.2]

4. Secondary Outcome: Progression Free Survival (PFS) Time as Measured From Start of 1st Line Platinum Therapy
Description: as for outcome 3
Time Frame: Up to two years post treatment discontinuation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
months | 9.9 [8.3 to 11.3]

5. Secondary Outcome: Overall Survival (OS) Time as Measured From Treatment Start
Time Frame: Up to two years post treatment discontinuation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
months | 15.9 [9.8 to 19.4]

6. Secondary Outcome: Overall Survival (OS) Time as Measured From Start of 1st Line Platinum Therapy
Time Frame: Up to two years post treatment discontinuation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rucaparib and Nivolumab
Number analyzed (Participants) | 31
months | 21.4 [14.8 to 25.7]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 5 year period.
Description: Adverse Events and All-Cause Mortality will be evaluated with secondary endpoints as data is still being collected.
Arm/Group | Rucaparib and Nivolumab
All-Cause Mortality (participants affected / at risk) | 26/31
Serious Adverse Events (participants affected / at risk) | 17/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib and Nivolumab (N=31)
Upper respiratory infection (Infections and infestations) | 1 (1)
Abdominal pain (General disorders) | 3 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) — Disease Progression
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 2 (2)
Biliary tract infection (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Disease Progression
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — COVID-19
Blood bilirubin increased (Investigations) | 2 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Post procedure discomfort
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rucaparib and Nivolumab (N=31)
Alkaline phosphatase increased (Investigations) | 2 (15)
Aspartate aminotransferase increased (Investigations) | 2 (24)
Bloating (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Dizziness (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (23)
Headache (General disorders) | 2 (3)
Hyperglycemia (Investigations) | 4 (19)
Hypocalcemia (Investigations) | 3 (7)
Hypotension (Vascular disorders) | 3 (4)
Lymphocyte count decreased (Investigations) | 3 (11)
Nausea (Gastrointestinal disorders) | 2 (12)
Neutrophil count decreased (Investigations) | 2 (17)
Photosensitivity (Eye disorders) | 2 (2)
Platelet count decreased (Investigations) | 3 (30)
Pruritus (Investigations) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT03639935/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT03639935/ICF_001.pdf